CLINICAL TRIAL: NCT05099276
Title: Extended Postoperative Tranexamic Acid Use in Primary Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial
Brief Title: Extended Postoperative Oral Tranexamic Acid in Knee Replacement
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Marcus C. Ford, Research Manager, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-08313-FB
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis; Blood Loss; Pain, Postoperative
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage; Pain, Postoperative | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Both oral TXA and oral placebo will be distributed to subjects in bottle marked with subject name and instructions for use following discharge from PACU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral TXA (Experimental): 1,950 mg oral tranexmic acid (three capsules of 650 mg) administered in post-anesthesia care, postop day one and postop day two. Compounded by registered pharmacist and labeled with subject name and instructions for use.
  Interventions: Drug: Tranexamic Acid Pill
- Oral placebo (Placebo Comparator): Three capsules of cellulose administered in post-anesthesia care, postop day one and postop day two. Compounded by registered pharmacist and labeled with subject name and instructions for use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid Pill — 1950 mg tranexamic acid (three capsules) given in post-anesthesia room and three capsules for postop day one and three capsules for postop day two
  Arms: Oral TXA
Drug: Placebo — Three capsules of cellulose given in post-anesthesia room and three capsules for postop cay one and three capsules for postop day two
  Arms: Oral placebo

SUMMARY:
A comparison of outcomes between use of oral tranexamic acid as compared to oral placebo in the first days after total knee replacement will be made to determine impact on clinical indications and patient reported outcomes.

DETAILED DESCRIPTION:
Significant blood loss occurs during total knee arthroplasty (TKA) which can lead to adverse outcomes including need for blood transfusion as well as increased local tissue swelling and ecchymosis which can inhibit post-operative recovery. Tranexamic acid (TXA), an inhibitor of fibrinolysis, has been shown to be a safe and effective drug for reducing blood loss during and after TKA. The use of TXA intraoperatively has been associated with higher postoperative hemoglobin levels and a reduction in postoperative blood transfusion rates. Administration of TXA in TKA has also been associated with improved clinical outcome measures including decreased rate of periprosthetic joint infection, decreased length of stay, and increased postoperative range of motion and early ambulation distances. However, there remains a wide variance in the route of administration, dosage, and timing of TXA use among treatment protocols in TKA. Previous studies have evaluated outcomes with the addition of post-operative TXA dosing to standard pre-operative and intra-operative intravenous (IV) doses. This study will investigate patient outcomes following a standardized post-operative oral TXA protocol as compared to oral placebo for three doses over day of surgery, postop day one and postop day two after TKA.

Following written consent documentation, Subjects will be randomized and blinded to randomization assignment until completion of study to either the oral TXA group or oral placebo group. The study medication will be distributed with the Subject's name with instructions for use in the post-anesthesia unit (PACU). The first dose will be administered in PACU with subsequent doses to be taken at home on postop day one and postop day two. TKA will be completed in an ambulatory surgery center with discharge same day of surgery to home.

Outcome measures include: Hemoglobin, visual analog score, KOOS Jr (Knee injury and osteoarthritis outcome score), range of motion, and incidence of treatment-emergent adverse event at postoperative (POD) day 3, POD week 2, POD week 6, and POD week 12. KOOS Jr. will be collected at one year post-op.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement in ambulatory setting
* Willing to participate
* Physical therapy on site at Campbell Clinic Wolf River
* Fluent in oral and written English

Exclusion Criteria:

* Unwilling to participate
* Revision total knee replacement
* Preoperative use of anticoagulants other than 81 mg aspirin
* Previous history of thromboembolic event
* Previous history of cancer other than non-melanoma skin cancers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | preoperative
  Hemoglobin enables red cells to transport oxygen and carbon dioxide in the blood and is measured in grams per deciliter with normal ranges of 12.0 to 17.5
Hemoglobin level | postoperative hour 3
  Hemoglobin enables red cells to transport oxygen and carbon dioxide in the blood and is measured in grams per deciliter with normal ranges of 12.0 to 17.5
Hemoglobin level | postoperative day 3
  Hemoglobin enables red cells to transport oxygen and carbon dioxide in the blood and is measured in grams per deciliter with normal ranges of 12.0 to 17.5
Hemoglobin level | postoperative week 2
  Hemoglobin enables red cells to transport oxygen and carbon dioxide in the blood and is measured in grams per deciliter with normal ranges of 12.0 to 17.5

SECONDARY OUTCOMES:
Visual Analog Score | preoperative
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | postoperative hour 3
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | postoperative week 2
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | postoperative week 6
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | postoperative week 12
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
KOOS Jr Score | preoperative
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
KOOS Jr Score | postoperative day 3
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
KOOS Jr Score | postoperative week 2
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
KOOS Jr Score | postoperative week 6
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
KOOS Jr Score | postoperative week 12
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
KOOS Jr Score | postoperative one year
  Patient reported outcome of how the knee feels from 0 to one 100 where 0 represents extreme problems and 100 represents no problems
range of motion of knee | preoperative
  clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion
range of motion of knee | postoperative day 3
  clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion
range of motion of knee | postoperative week 2
  clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion
range of motion of knee | postoperative week 6
  clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion
range of motion of knee | postoperative week 12
  clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion

OTHER OUTCOMES:
Incidence of treatment-emergent adverse event | postoperative day 3
  monitoring for safety events
Incidence of treatment-emergent adverse event | postoperative week 2
  monitoring for safety events
Incidence of treatment-emergent adverse event | postoperative week 6
  monitoring for safety events
Incidence of treatment-emergent adverse event | postoperative week 12
  monitoring for safety events

CONTACTS AND LOCATIONS:
Overall Officials: Marcus C Ford, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Shores P, Mullen K, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. The Safety of Tranexamic Acid in Total Joint Arthroplasty: A Direct Meta-Analysis. J Arthroplasty. 2018 Oct;33(10):3070-3082.e1. doi: 10.1016/j.arth.2018.03.031. Epub 2018 Mar 22. PMID 29699826
- [Result] Rutherford RW, Jennings JM, Dennis DA. Enhancing Recovery After Total Knee Arthroplasty. Orthop Clin North Am. 2017 Oct;48(4):391-400. doi: 10.1016/j.ocl.2017.05.002. Epub 2017 Aug 8. PMID 28870300
- [Result] Prasad N, Padmanabhan V, Mullaji A. Blood loss in total knee arthroplasty: an analysis of risk factors. Int Orthop. 2007 Feb;31(1):39-44. doi: 10.1007/s00264-006-0096-9. Epub 2006 Mar 28. PMID 16568327
- [Result] Kim JK, Park JY, Lee DY, Ro DH, Han HS, Lee MC. Optimal dose of topical tranexamic acid considering efficacy and safety in total knee arthroplasty: a randomized controlled study. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3409-3417. doi: 10.1007/s00167-020-06241-9. Epub 2020 Aug 31. PMID 32869124
- [Result] Wu C, Tan C, Wang L. Higher doses of topical tranexamic acid safely improves immediate functional outcomes and reduces transfusion requirement in total knee arthroplasty. Arch Orthop Trauma Surg. 2020 Dec;140(12):2071-2075. doi: 10.1007/s00402-020-03591-4. Epub 2020 Aug 29. PMID 32862267
- [Result] Drain NP, Gobao VC, Bertolini DM, Smith C, Shah NB, Rothenberger SD, Dombrowski ME, O'Malley MJ, Klatt BA, Hamlin BR, Urish KL. Administration of Tranexamic Acid Improves Long-Term Outcomes in Total Knee Arthroplasty. J Arthroplasty. 2020 Jun;35(6S):S201-S206. doi: 10.1016/j.arth.2020.02.047. Epub 2020 Mar 4. PMID 32209286
- [Result] Grosso MJ, Trofa DP, Danoff JR, Hickernell TR, Murtaugh T, Lakra A, Geller JA. Tranexamic acid increases early perioperative functional outcomes after total knee arthroplasty. Arthroplast Today. 2017 Jun 29;4(1):74-77. doi: 10.1016/j.artd.2017.05.009. eCollection 2018 Mar. PMID 29560399
- [Result] Torkaman A, Rostami A, Sarshar MR, Akbari Aghdam H, Motaghi P, Yazdi H. The Efficacy of Intravenous Versus Topical Use of Tranexamic Acid in Reducing Blood Loss after Primary Total Knee Arthroplasty: A Randomized Clinical Trial. Arch Bone Jt Surg. 2020 May;8(3):363-367. doi: 10.22038/abjs.2020.40528.2099. PMID 32766393
- [Result] Lei Y, Xie J, Huang Q, Huang W, Pei F. Additional benefits of multiple-dose tranexamic acid to anti-fibrinolysis and anti-inflammation in total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2020 Aug;140(8):1087-1095. doi: 10.1007/s00402-020-03442-2. Epub 2020 Apr 6. PMID 32253548
- [Result] Pavenski K, Ward SE, Hare GMT, Freedman J, Pulendrarajah R, Pirani RA, Sheppard N, Vance C, White A, Lo N, Waddell JP, Ho A, Schemitsch EH, Kataoka M, Bogoch ER, Saini K, David Mazer C, Baker JE. A rationale for universal tranexamic acid in major joint arthroplasty: overall efficacy and impact of risk factors for transfusion. Transfusion. 2019 Jan;59(1):207-216. doi: 10.1111/trf.14995. Epub 2018 Nov 1. PMID 30383292
- [Result] Luo ZY, Wang HY, Wang D, Zhou K, Pei FX, Zhou ZK. Oral vs Intravenous vs Topical Tranexamic Acid in Primary Hip Arthroplasty: A Prospective, Randomized, Double-Blind, Controlled Study. J Arthroplasty. 2018 Mar;33(3):786-793. doi: 10.1016/j.arth.2017.09.062. Epub 2017 Oct 6. PMID 29107495
- [Result] Wang HY, Wang L, Luo ZY, Wang D, Tang X, Zhou ZK, Pei FX. Intravenous and subsequent long-term oral tranexamic acid in enhanced-recovery primary total knee arthroplasty without the application of a tourniquet: a randomized placebo-controlled trial. BMC Musculoskelet Disord. 2019 Oct 25;20(1):478. doi: 10.1186/s12891-019-2885-5. PMID 31653221
- [Result] Wang D, Wang HY, Luo ZY, Meng WK, Pei FX, Li Q, Zhou ZK, Zeng WN. Blood-conserving efficacy of multiple doses of oral tranexamic acid associated with an enhanced-recovery programme in primary total knee arthroplasty: a randomized controlled trial. Bone Joint J. 2018 Aug;100-B(8):1025-1032. doi: 10.1302/0301-620X.100B8.BJJ-2017-1598.R1. PMID 30062946